CLINICAL TRIAL: NCT05659225
Title: Telemedicine System and Intelligent Monitoring System Construction of Pediatric Asthma Based on the Electronic Stethoscope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SCMCIRB-YJ2022002
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-11

CONDITIONS: Asthma
Keywords: Pediatric; Asthma Control; Electronic Stethoscope
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electronic stethoscope group (Other): During the study, subjects who diagnosed as asthma according to "Guideline for the diagnosis and optimal management of asthma in children" will be assigned to the control group and the electronic stethoscope group, and receive 12 months standard treatment, prescribed by the investigators according to "Guideline for the diagnosis and optimal management of asthma in children". The patient's caregiver will be instructed to use an electronic stethoscope to coordinate treatment and complete follow-up.
  Interventions: Device: Electronic Stethoscope; Other: Standard treatment according to GINA(2019)
- control group (Other): During the study, subjects who diagnosed as asthma according to "Guideline for the diagnosis and optimal management of asthma in children" will be assigned to the control group and the electronic stethoscope group, and receive 12 months standard treatment, prescribed by the investigators according to "Guideline for the diagnosis and optimal management of asthma in children".
  Interventions: Other: Standard treatment according to GINA(2019)

INTERVENTIONS:
Device: Electronic Stethoscope — Subjects diagnosed as pediatric asthma at Shanghai Children's Medical Center will be consecutively screened and eligible patients will be recruited (enrolment visit, V1). The subject will be assigned to the control group and the electronic stethoscope group and complete their future onsite visits (V2-V5) at Shanghai Children's Medical Center. The patient's caregiver who was assigned to the electronic stethoscope group will be instructed to install the electronic stethoscope developed by our team and its accessories, then they will be trained by investigators on how to use the electronic stethoscope.
  Other Names: study-specified asthma device program
  Arms: electronic stethoscope group
Other: Standard treatment according to GINA(2019) — Subjects diagnosed as pediatric asthma at Shanghai Children's Medical Center will be consecutively screened and eligible patients will be recruited (enrolment visit, V1). The subject will be assigned to the control group and the electronic stethoscope group and complete their future onsite visits (V2-V5) at Shanghai Children's Medical Center. The patient's caregiver who was assigned to the control group will receieve standard treatment according to GINA(2019).

SUMMARY:
The purpose of this study is to retrofit the existing electronic stethoscope, improve the quality and efficiency of signal acquisition and the intelligent degree of information processing, decrease the manual action of electronic stethoscopes implemented by parents of asthma children, simplify the process of data transfer and the user's operational cost using signal processing, artificial intelligence technology, thus decreasing the feedback cycle between patients and clinicians. Eventually, we will construct an intelligent monitoring system based on the modified electronic stethoscope and explore the interactive remote management approaches on children's asthma at the same time, thus achieving revolutionized remote management of asthma.

DETAILED DESCRIPTION:
(1) The design of hardware and software of the intelligent electronic stethoscope This project will optimize and develop the software and hardware equipment of electronic stethoscope according to the shortcomings of existing electronic stethoscopes.

1. Get high-quality breath sound data through integrated ECG sensor and algorithms for denoising and the separation of heart sound and lung sound
2. Develop algorithms and corresponding frameworks for visualization of breath sounds and mining of key information
3. Develop algorithms for automatic recognition of abnormal breath sounds
4. Transfer breath sound data efficiently and reliably based on the encoding-decoding architecture
5. Optimize the breath sound data transmission process
6. Construct the remote diagnosis and treatment methods and monitoring system for childhood asthma preliminary

(2) The effect of telemedicine system and intelligent monitoring system based on intelligent stethoscope on children with asthma Subjects diagnosed as pediatric asthma at Shanghai Children's Medical Center will be consecutively screened and eligible patients will be recruited. For each enrolled patient, basic information as well as baseline medical condition will be collected by the investigators. The subject will be randomly assigned to the control group and the electronic stethoscope group. The patient's caregiver who was assigned to the electronic stethoscope group will be instructed to install the electronic stethoscope developed by our team and its accessories, then they will be trained by investigators on how to use the electronic stethoscope.

During the study, patients will receive 12 months standard treatment, prescribed by the investigators according to "Guideline for the diagnosis and optimal management of asthma in children". If patients develop upper respiratory tract symptoms without fever, the investigator will give corresponding guidance to the control group and the electronic stethoscope group. If fever develops, it is recommended that patients directly go to the emergency department.

All patients' caregiver will be prompted to finish the test for respiratory and asthma control in kids (TRACK) every month. Patient's caregiver assigned to the electronic stethoscope group will also need to complete the collection, data upload and sharing of patient's breath sounds at least once a month to confirm that the electronic stethoscope is worked correctly.

After enrollment, patients will be requested to visit Shanghai Children's Medical Center at month 3, 6, 9, 12. During each onsite visit, subjects will receive lung function (≥4 years) and FENO tests and fill out the questionnaire regarding the number of asthma-related outpatient emergency department visits, asthma-related hospitalizations, SABA and systemic glucocorticoid use, missed work and school misses, and asthma-related medical expenses in the past 3 months. At 6- and 12-month's visit, pediatric asthma caregiver's quality of Life questionnaire (PACQLQ) needs to be completed at the same time.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as asthma according to "Guideline for the diagnosis and optimal management of asthma in children" in the respiratory clinic of Shanghai Children's Medical Center from January 2023 to January 2025
2. Out-patient, female or male, 3 years old≤ age < 6 years old
3. long-term maintenance therapy with inhaled glucocorticoids or concomitant leukotriene receptor antagonists
4. Equipped with a household atomizer or spacer, it can afford the inhalation therapy of short-acting β2 receptor agonists (SABA) at home
5. The subjects or subjects' caregiver must have a smart phone with Android or Harmony system at their disposal
6. The guardian agrees to participate in the study and signs the informed consent form

Exclusion Criteria:

1. Acute exacerbation of asthma 30 days before enrollment (receive short-term prednisone treatment, emergency department visit or hospitalization due to acute asthma attacks)
2. Other chronic lung diseases, cardiovascular diseases, blood system diseases, immunodeficiency diseases, neurological diseases, genetic or chromosomal abnormalities and other underlying diseases
3. Patients or their caregivers can't complete the collection of breath sound

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
visits of asthma-related unplanned emergency department | 1 year
  Subjects will fill out a questionnaire to provide the number of unscheduled emergency department visits related to asthma (except for routine asthma follow-up visits every 3 months).

SECONDARY OUTCOMES:
asthma control | 1 year
  The patients' caregiver will be prompted to fill out an asthma control questionnaire every month. This questionnaire contains questions regarding renewal of prescription, control status and asthma attack.
adherence to asthma treatment | 1 year
  Patients' adherence will be assessed by investigator through questionnaire.

OTHER OUTCOMES:
SABA use | 1 year
  Number of days and total amount of SABA use will be collected by investigator through questionnaire.
systemic corticosteroid use | 1 year
  Days of systemic corticosteroid use will be counted by investigator through questionnaire.
lung function | 1 year
  Subjects (equal or older than 4 years) will receive PEF (Peak expiratory flow, L/min) tests for evaluation of lung function.
FENO tests | 1 year
  Subjects will receive FENO (Fractional exhaled nitric oxide, parts per billion, ppb) tests for evaluation of lung inflammation level.
Asthma-related medical expenses | 1 year
  Asthma-related medical expenses will be counted by investigator through questionnaire.
Asthma-related hospitalizations | 1 year
  Number of asthma-related hospitalizations will be collected by investigator through questionnaire.
Missed school and parents missed work | 1 year
  Number of missed school and parents missed work will be collected by investigator through questionnaire.
Patients' and caregivers' quality of life | 1 year
  Patients' and caregivers' quality of life will be evaluated by investigator through questionnaire.
Caregivers' satisfaction degree with electronic stethoscopes | 1 year
  Caregivers' satisfaction degree with electronic stethoscopes will be assessed by investigators through questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Yin, PhD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China